CLINICAL TRIAL: NCT00596596
Title: A Double-Blind, Placebo-Controlled, Dose-Finding Trial to Evaluate the Efficacy and Safety of Prucalopride (R093877) in Subjects With Chronic Idiopathic Constipation
Brief Title: Trial to Evaluate the Efficacy and Safety of R093877 in Patients With Chronic Idiopathic Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Movetis (Industry)
Responsible Party: Renate Specht Gryp, Movetis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRU-USA-3
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-01

CONDITIONS: Constipation
Keywords: Constipation; prucalopride
MeSH Terms: conditions — Constipation | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Active Comparator): 0,5 mg prucalopride
  Interventions: Drug: prucalopride
- 2 (Active Comparator): 1 mg prucalopride
  Interventions: Drug: prucalopride
- 3 (Active Comparator): 2 mg prucalopride
  Interventions: Drug: 2 mg prucalopride
- 5 (Placebo Comparator): Placebo arm
  Interventions: Other: Placebo
- 4 (Active Comparator): 4 mg prucalopride
  Interventions: Drug: 4 mg prucalopride

INTERVENTIONS:
Drug: prucalopride — 0,5 mg once daily
  Other Names: Resolor
  Arms: 1
Drug: prucalopride — 1 mg once daily
  Other Names: Resolor
  Arms: 2
Drug: 2 mg prucalopride — 2 mg once daily
  Other Names: Resolor
  Arms: 3
Drug: 4 mg prucalopride — 4 mg once daily
  Other Names: Resolor
  Arms: 4
Other: Placebo — placebo once daily
  Arms: 5

SUMMARY:
The purpose of the study is to determine whether prucalopride is safe and effective in patients with chronic idiopathic constipation.

Hypothesis:

At all doses administered prucalopride given once daily for 4 weeks is safe and well tolerated in patients with chronic idiopathic constipation.

DETAILED DESCRIPTION:
This was a double-blind, placebo-controlled, randomized, parallel group, multicentre, Phase II, dose comparison trial, in which 313 subjects, with a history of chronic idiopathic constipation were enrolled. The trial was conducted in three phases:

1. a 4-week drug-free run-in phase,
2. a 4-week double-blind (DB) phase during which subjects were treated with R093877 (0.5 mg, 1 mg, 2 mg, or 4 mg capsule) or matching placebo once daily, prior to breakfast,
3. a 4-week drug-free run-out phase (RO).

To qualify for the run-in phase (Visit 1, Week 1) subjects had to have experienced, for at least 3 months, 2 or less spontaneous, bowel movements (SBM)/week with the occurrence of lumpy (scyballae) and/or hard stools, a sensation of incomplete evacuation for at least a quarter of their stools, or straining during defecation at least a quarter of the time.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female outsubjects between 18 and 70 years of age.
* Documented history of constipation. The subject reports 2 or less SCBM/week with the occurrence of one or more of the following for at least 3 months before selection visit:

  * lumpy (scyballae) and/or hard stools at least a quarter of the stools;
  * sensation of incomplete evacuation following at least a quarter of the stools; or
  * straining at defecation at least a quarter of the time.

These criteria were only applicable for spontaneous, complete bowel movements, i.e., not preceded within a period of 24 hours by the intake of a laxative agent.

* Normal inhibition pattern of the external anal sphincter during straining, i.e., relaxation of the m. puborectalis and a distal displacement of the rectal canal (digital examination and/or electromyographic and/or manometric evidence was acceptable).
* The subject's constipation was functional, i.e., idiopathic.
* Written informed consent, signed by the subject and/or legal guardian and by the investigator.
* Subject were available for follow-up during the trial period, as determined in the protocol.

Exclusion Criteria:

* Subjects in whom constipation was thought to have been drug-induced.
* Subject who suffered from types/causes of constipation other than idiopathic constipation, i.e.,presence of secondary causes of constipation including:

  * Endocrine disorders
  * Metabolic disorders
  * Neurologic disorders including:
* Irritable bowel syndrome.
* Subjects with congenital megacolon/megarectum or a diagnosis or pseudo-obstruction.
* History of previous abdominal surgery (excluding hysterectomy, surgery for Meckel's diverticle,appendectomy, cholecystectomy, inguinal hernia repair, splenectomy, nephrectomy, fundoplication)thought to have been the primary cause of constipation.
* Known or suspected organic disorders of the large bowel (i.e., obstruction, carcinoma, or inflammatory bowel disease). -Subjects with active proctological conditions thought to have been responsible for the constipation.
* Subjects with ECG abnormalities including:

  * 2nd or 3rd degree AV block;
  * prolonged QTc intervals (> 460 msec); or
  * bradycardia (< or equal to 60 bpm).
* Subjects who were receiving concomitant medication which could cause QT prolongation
* Subjects on potassium-wasting diuretics.
* Subjects with known illnesses or conditions such as:

  * severe cardiovascular or lung disease,
  * neurologic or psychiatric disorders (including active alcohol or drug abuse),
  * cancer,
  * AIDS, or
  * other gastrointestinal or endocrine disorders.
* Subjects with impaired renal function
* Subjects with a serum amylase, AST (SGOT), or ALT (SGPT) concentration >2 times the normal limit.
* Subjects with clinically significant abnormalities of hematology, urinalysis or blood chemistry.
* Females of childbearing potential without adequate contraceptive protection during the trial. Oral
* Females who were pregnant or lactating.
* Subjects who received an investigational drug in the 30 days preceding the run-in phase of this trial.
* Subjects who were unable or unwilling to return for required follow-up visits.
* Subjects whose reliability or physical state hindered adequate participation in a clinical trial.
* Subjects who had polyps discovered during the screening colonoscopy that were untreated (i.e., by polypectomy). Subjects who had polyps during the screening colonoscopy that were treated by polypectomy were allowed to enter the trial after the 4-week healing period. Any subject with polyp(s)documented to contain an invasive carcinoma (Duke's B or greater) was excluded from this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 1996-09; Primary Completion 1997-06 (Actual); Study Completion 1997-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the optimal dose of R093877 for the treatment of chronic idiopathic constipation by comparing the efficacy and safety of 0.5 mg, 1 mg, 2 mg, and 4 mg of R093877 versus placebo given orally once daily for 4 weeks. | 4 weeks

SECONDARY OUTCOMES:
Evaluation of the effects of R093877 on symptoms associated with idiopathic constipation | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Trent Nichols, MD, Principal Investigator — Hanover General Hospital

REFERENCES:
- [Derived] Emmanuel A, Cools M, Vandeplassche L, Kerstens R. Prucalopride improves bowel function and colonic transit time in patients with chronic constipation: an integrated analysis. Am J Gastroenterol. 2014 Jun;109(6):887-94. doi: 10.1038/ajg.2014.74. Epub 2014 Apr 15. PMID 24732867